CLINICAL TRIAL: NCT05538598
Title: Effect of Intramuscular Dry Needling on Soft Tissue Stiffness and Pressure-pain Thresholds
Brief Title: Dry Needling and Muscle Stiffness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research personnel.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Koehle, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H22-01852
Record Dates: First submitted 2022-09-07; First posted 2022-09-14 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Muscle Tightness

STUDY DESIGN:
Intervention Model Description: Repeated measures design with pre-post measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intramuscular Dry Needling (Experimental): IMDN will be performed at the sacral multifidus and fibularis longus muscles.
  Interventions: Procedure: Intramuscular Dry Needling

INTERVENTIONS:
Procedure: Intramuscular Dry Needling — The insertion of thin monofilament needles (without injectate) into a tight band of muscle. The needles will be inserted into the muscle for ~10 seconds.

SUMMARY:
The goal of this study is to investigate the effect of intramuscular dry needling (IMDN) on muscle stiffness and pain. Research has suggested that IMDN can reduce muscle stiffness in needled areas. As well, IMDN may reduce mechanical pain sensitivity experienced by individuals.

IMDN will be performed at several anatomical locations. Muscle stiffness will be measured with a handheld probe, which measures contact force and displacement of soft tissue. Pressure-pain thresholds (PPT) will be discovered at each region of interest. Stiffness and pressure-pain thresholds will be collected before and after IMDN. The data collected from this research is important to understand the mechanism of IMDN and its relationship to pain.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* pain-free in your lower back and lower legs

Exclusion Criteria:

* unable to communicate in English
* surgery of any kind in the lumbar spine or lower legs.
* participants with a skin condition that does not allow for hypoallergenic tape to be attached to their skin.
* have a BMI>25
* unable to hold your breath for 20 seconds
* contraindications to dry needling, i.e. pregnancy; fever or infection that is in your bloodstream; unstable compromised immune system; unstable bleeding disorders; presence at the site of DN of infection, an open wound , a burn, cellulitis, or an undiagnosed lump; post- mastectomy/lymph node removal in the affected limb; post-major surgery (3-6 month time period); presence of metal or plastic implant; absent sensation in area of planned DN; post-bacterial endocarditis or heart valve conditions/replacement without medical clearance for DN from medical doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effective stiffness of soft tissue | Within 10 minutes of intervention
  Force-displacement data is collected while deforming the soft tissue at the skin surface with a non-invasive handheld probe. The effective stiffness is a summary of the deformation behavior of the soft tissue. It is estimated using the force-displacement data as an input to the incompressible isotropic hyperelastic Ogden model. A higher value indicates that the soft tissue is stiffer than a lower value.
Pressure-pain threshold | Within 10 minutes of intervention
  The measured pressure at the moment the perception of pressure turns into pain

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koehle, MD, PhD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No